CLINICAL TRIAL: NCT03106051
Title: Long-term Documentation on the Use of Apremilast in Patients With Psoriatic Arthritis in Practice Conditions
Brief Title: Study of Apremilast Use in Patients With Psoriatic Arthritic in Practice Conditions
Acronym: LAPIS-PsA
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-10004-PSA-008
Record Dates: First submitted 2017-03-17; First posted 2017-04-10 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Arthritis, Psoriatic
Keywords: Arthritis; Psoriatic; Observational; Apremilast
MeSH Terms: conditions — Arthritis, Psoriatic; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with active psoriatic arthritis: Patients who suffer from active psoriatic arthritis with at least moderate disease corresponding to a PGA of ≥2

SUMMARY:
A total of approximately 500 patients with active psoriatic arthritis in an estimated 80 to 100 trial centers are to be enrolled. Selection of centers will be made by the sponsor's medical section. To increase the quality of the data and to reduce distribution of the data collected, centers to be included will be those which can enroll at least 5 patients. Care will be taken to ensure a balanced regional distribution. The proposed observation period for the trial is approx. 52 weeks per patient. Estimated patient enrolment is also 52 weeks. The duration of the follow-up period will be extended from approx. 52 weeks to approx. 100 weeks to gain further information about the long-term use of Otezla®. For this extension of the follow-up period 2 new visits (visits 6 and 7) are proposed.Thus, proposed duration from first patient in (FPI) to last patient out (LPO) is 36 months-

ELIGIBILITY:
Inclusion Criteria:

* The decision to treat with Otezla® has been made independently before inclusion in this study
* Patient age ≥ 18 years
* Existing diagnosis of active psoriatic arthritis
* At least moderately severe psoriatic arthritis (Physician's Global Assessment (PGA) scale ≥ 2)
* Insufficient response or intolerance to previous Disease-Modifying Anti-Rheumatic Drug (DMARD) treatment (disease modifying anti-rheumatic drugs)
* A written informed consent statement by the patient permitting data collection, evaluation, storage and transfer

Exclusion Criteria:

* Pregnancy
* Hypersensitivity to apremilast or one of the other ingredients in the film tablets
* Other criteria according to the summary of product characteristics Breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Overall approx. 500 patients with active psoriatic arthritis are to be enrolled. Inclusion and exclusion criteria derive from the current Otezla® summary of product characteristics and the criteria.
Sampling Method: Non-Probability Sample
Enrollment: 526 (Actual)
Dates: Start 2016-02-18 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with an improvement of ≥ 1 points on the Physician's Global Assessment (PGA) scale on visit 3 compared to baseline on the Physician's Global Assessment scale (PGA; scale from 0-4) | Up to approximately 7 months
  Physician's global assessment (PGA) will be measured on a VAS scale ranging from 0 to 4. Primary endpoint is the percentage of patients with an improvement of minimum 1 point on this VAS scale after about 6 months (visit 3)

SECONDARY OUTCOMES:
Percentage of patients with an improvement of ≥ 1 points on the Patient Global Assessment (PaGA) scale on visits 1 to 7 compared to baseline | Up to approximately 104 weeks
  Patient Global Assessment will be measured on a VAS scale ranging from 0 to 5. The percentage of patients with an improvement of minimum 1 point will be measured throughout the study.
Percentage of patients with an improvement of ≥ 1 points on the Physician's Global Assessment (PGA) scale on visits 1, 2, 4, 5, 6, 7 compared to baseline | Up to approximately 104 weeks
  Additionally to the primary endpoint the improvement of the PGA of minimum 1 point will be measured throughout the study.
Efficacy of the treatment with regard to rheumatic changes measured with Tender Joint Count (TJC) on visits 1 to 7 compared to baseline | Up to approximately 104 weeks
  Tender Joint Count will be measured throughout the study and compared to baseline.
Efficacy of the treatment with regard to rheumatic changes measured with Swollen Joint Count (SJC) on visits 1 to 7 compared to baseline | Up to approximately 104 weeks
  Swollen Joint Count will be measured throughout the study and compared to baseline.
Efficacy of the treatment with regard to rheumatic changes measured with Visual Analog Scale (VAS) on visits 1 to 7 compared to baseline- Pain | Up to approximately 104 weeks
  Visual Analog Scale; scale from 0-100 to question how the patient feels subjectively about their pain (0 = no pain, 100 = worst imaginable pain)
Psoriatic arthritis Impact of Disease (PsAID) questionnaire on visits 1, 2, 3, 5 and 7 compared to baseline | Up to approximately 104 weeks
  Improvement of the Impact of Disease (PsAID) will be measured during visit 1, 2 and 5 and compared to baseline
Hannover Functional Ability Questionnaire (FFbH) on visits 1, 2, 3, 5 and 7 compared to baseline | Up to approximately 104 weeks
  Composite score to measure functional improvement will be measured during visits 1, 2 and 5 and compared to baseline
Patient Preference Questionnaire (PPQ) on visits 3, 5 and 7 | Up to approximately 104 weeks
  The therapy preference of the patient will be measured compared to his previous systemic therapy
Assessment of psoriatic skin changes (Body Surface Area, BSA) on visits 1 to 7 | Up to approximately 104 weeks
  Extension of the psoriatic plaques will be measured by body surface area (BSA) throughout the study
Adverse Events (AEs) | Up to approximately 104 weeks
  Number of subjects with adverse events
Efficacy of the treatment with regard to rheumatic changes measured with Visual Analog Scale (VAS) on visits 1 to 7 compared to baseline- Enthesitis | Up to approximately 104 weeks
  Visual Analog Scale; scale from 0-100 to question how the patient feels subjectively about their enthesitis (0 = no enthesitis, 100 = worst imaginable enthesitis)
Efficacy of the treatment with regard to rheumatic changes measured with Visual Analog Scale (VAS) on visits 1 to 7 compared to baseline- Joints | Up to approximately 104 weeks
  Visual Analog Scale; scale from 0-100 to question how the patient feels subjectively about their joints (0 = no affected joints, 100 = heavily affected joints)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- Germany (2):
  - Rheumatology at Struenseehaus, Altona, Hamburg
  - Klinikum Stephansplatz, Hamburg

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com